CLINICAL TRIAL: NCT05014737
Title: External Validation of Two Models to Predict Postoperative Nausea and Vomiting (PONV) in Patients With Liver Cancer in Chinese Hospital Setting
Brief Title: External Validation of the Apfel Risk Score and Koivuranta Score to Predict Postoperative Nausea and Vomiting in Patients With Liver Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2020-347
Record Dates: First submitted 2021-08-17; First posted 2021-08-20 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Nausea and Vomiting; Hepatobiliary Surgery; Prediction Model
Keywords: Postoperative Nausea and Vomiting; hepatobiliary surgery; assessment tool
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with low risk of PONV
- Patients with high risk of PONV
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is an abservational study and no intervention will be involved
  Groups: Patients with high risk of PONV

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common complication among surgical patients. The incidence ranging from 20% to 50% depends on different population studied. Clinical practice guidelines recommend routine PONV screening before surgery using the Apfel simplified risk score OR Koivuranta score. However, these two scores haven't been translated into Chinese version and tested for psychometric qualities. Therefore, this study aim to externally validate two PONV prediction models in the Chinese hospital setting for PONV assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving hepatobiliary surgery

Exclusion Criteria:

* patients receiving chemothreapy；patients with cognitive disorders; patients unwilling to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving hepatobiliary surgery will be consectively invited, and PONV will be assessed within 24 hours after surgery．
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 24 hours after surgery
  Postoperative nausea will be assessed at 24 hours after surgery on an 11-point numeric scale (0 -10) by a trained nurse. Patients will be asked to respond to the question, "Have you felt nauseated since your discharge from the postanesthetic care unit and if so, what would be the average level of nausea you have felt until now on a 0 to 10 scale?". Patients will be considered nauseated if postoperative nausea is reported to be greater than zero on the 11-point scale with the question. For the same intervals the number of episodes of postoperative vomiting will be recorded. Again, patients will be considered to have vomited if postoperative vomiting occurs at least once within 24 hours. Patients who have either postoperative nausea or postoperative vomiting in 24h will be considered to have PONV.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available when asked with reasonable reasons.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code